CLINICAL TRIAL: NCT04432948
Title: Maternal Psychological Implications of Covid-19 Pandemic and Possible Effect on Anaesthetic Management.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: General and Maternity Hospital of Athens Elena Venizelou (Other)
Responsible Party: Principal Investigator, GEORGIA MICHA, Anesthesiologist MD, MSc, PhD, General and Maternity Hospital of Athens Elena Venizelou
Other Study IDs: Maternal Covid 19
Record Dates: First submitted 2020-06-14; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Covid-19; Maternal Psychological Distress; Anesthesia
Keywords: Covid-19; Psychological Distress; Maternal; Anaesthesia
MeSH Terms: conditions — COVID-19 | interventions — Patient Health Questionnaire

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Maternal Group: Pregnant women administered into a maternity public hospital in labour (vaginal delivery, caesarean section)
  Interventions: Other: PHQ-9 Depression Scale; Other: GAD-7 General anxiety disorder scale; Other: 38-questions questionnaire

INTERVENTIONS:
Other: PHQ-9 Depression Scale — It involves a 9-question scale that detects depression
Other: GAD-7 General anxiety disorder scale — It involves a 7-question scale that detects general anxiety disorder
Other: 38-questions questionnaire — It involves a 38 question questionnaire that aims to detect any association between the Covid-19 pandemic, the psychological impllications and anaesthetic practice

SUMMARY:
The aim of this study is to assess the maternal psychological implication of the novel coronavirus COvid-19 pandemic. At the same time it will be evaluated whether there is an impact of these implications on the anaesthetic practice.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women over the age of 18 that present in labour (vaginal delivery or caesarean section)

Exclusion Criteria:

* psychiatric disorders
* drug abuse
* not eligible to read and write in Greek

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — maternity
Study Population: All women in labour that present into the maternity hospital from June-August 2020, during the Covid-19 pandemic
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Association between Covid-19 pandemic and maternal psychological distress | Pre-labour assessment
  Association between Covid-19 pandemic and maternal psychological distress assessed by 2 scales and one questionnaire

SECONDARY OUTCOMES:
Association between Covid-19 pandemic, maternal psychological distress and anaesthetic practice | Pre-labour assessment
  Association between Covid-19 pandemic and anaesthetic practice assessed by a 38 questions questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Georgia Micha, Dr, Principal Investigator — Elena Venizelou General and Maternity Hospital of Athens, Greece
Locations (1):
- "Elena Venizelou" General and Maternity Hospital of Athens, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Thapa SB, Mainali A, Schwank SE, Acharya G. Maternal mental health in the time of the COVID-19 pandemic. Acta Obstet Gynecol Scand. 2020 Jul;99(7):817-818. doi: 10.1111/aogs.13894. No abstract available. PMID 32374420